CLINICAL TRIAL: NCT05271786
Title: WEANING FROM TRACHEOSTOMY: A MULTICENTER, OBSERVATIONAL REVIEW OF PROCEDURES AND PROTOCOLS AND A RESTROSPECTIVE VALIDATION OF THE QSQ SCORING SYSTEM
Brief Title: WEANING FROM TRACHEOSTOMY
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Collaborators: Dejan Radovanovic (Unknown); Marina Gatti (Unknown); Michele Mondoni (Unknown); Stefano Centanni (Unknown); Frascesco Blasi (Unknown); Andrea Gramegna (Unknown); Fabiano Di Marco (Unknown); Stefano Aliberti (Unknown); Humanitas Research Hospital IRCCS, Rozzano-Milan (Other); Ca' Granda Policlinico Milano (Unknown); ASST Santi Paolo e Carlo (Other); Ospedale Luigi Sacco Milano (Unknown); Papa Giovanni XXIII Bergamo (Unknown)
Responsible Party: Principal Investigator, Pierachille Santus, MD, PhD, Professor, University of Milan
Other Study IDs: OR022022
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Tracheostomy Weaning; Tracheostomy Decannulation
Keywords: tracheostomy weaning; tracheostomy decannulation; Quantitative-Semi Quantitative - QSQ
MeSH Terms: interventions — Tracheostomy Decannulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- Tracheostomized patients: Patients who underwent percutaneous tracheostomy performed for any reason
  Interventions: Other: Decannulation

INTERVENTIONS:
Other: Decannulation — retrospective evaluation of decannulation

SUMMARY:
Tracheostomy is a very common surgical procedure performed in critically ill patients on invasive mechanical ventilation, and usually performed in difficult-to-wean patients and whn prolonged mechanical ventilation is required.

Weaning from the tracheostomy cannula (i.e. decannulation) represents one of the crucial steps in the post-acute respiratory management of these patients. Tracheostomy literature mainly focuses on the timing and technique of this procedure, but there is a lack of studies about decannulation and, currently, our knowledge is primarily based on expert opinion. The COVID-19 pandemic, due to the rapid increase in the number of patients exposed to prolonged mechanical ventilation, has stressed the need for objective parameters and shared standardized protocols to perform weaning from tracheostomy.

DETAILED DESCRIPTION:
The study will have two co-primary objectives:

1. To review and compare the standard operating procedures adopted for decannulation at a multicenter level.
2. To retrospectively validate a clinical score for weaning from trachesotomy (Quantitative-Semi Quantitative - QSQ) Secondary objectives will be: 1) to assess the presence of predictors of decannulation failure; 2) to investigate if timing of decannulation can influence the result of the tracheostomy weaning process, and 3) to possibly derive a novel clinical score and a shared protocol for decannulation.

The investigators will retrospectively collect data from patients who underwent a tracheostomy procedure and decannulation during their hospital stay since January 2017 until November 2021.

A digital dataset will be shared with the participating centers. The following variables will be collected: age, gender, comorbidities, reason and date of tracheostomy, technique used, type of cannula, variables associated with the weaning process (timing and type of caliber reduction, tube capping, assessment of airway patency by means of fiberoptic bronchoscopy, effectiveness of cough and swallowing, type and timing of change in respiratory support), level of consciousness, vital signs, arterial blood gas analysis and blood tests before and after decannulation, failure of decannulation and related complications. The dataset will be also designed to retrospectively validate the QsQ score, which is based on two main criteria (or quantitative parameters) and eight minor criteria (or semi-quantitative parameters).

Inclusion criteria

1. Patients >18 years old
2. Percutaneous tracheostomy performed for any reason
3. At least one decannulation attempt during the hospitalization period. Exclusion criteria

1. Patients with surgical/permanent tracheostomy (e.g. neuromuscular disorders needing long-term invasive mechanical ventilation) 2. Patients that underwent elective tracheostomy due to neck masses or tumors, in view of a surgical approach 3. Patients tracheostomized more than once

ELIGIBILITY:
Inclusion Criteria:

1. Patients >18 years old
2. Percutaneous tracheostomy
3. At least one decannulation attempt

Exclusion Criteria:

1. Surgical/permanent tracheostomy
2. Elective tracheostomy due to neck masses or tumors, in view of a surgical approach
3. Patients tracheostomized more than once

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent a tracheostomy procedure and decannulation during their hospital stay since January 2017 until November 2021.
Sampling Method: Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Standard procedures of decannulation | 5 years
  To review and compare the standard operating procedures adopted for decannulation at a multicenter level.
QSQ score | 5 years
  To retrospectively validate a clinical score for weaning from trachesotomy (Quantitative-Semi Quantitative - QSQ )

SECONDARY OUTCOMES:
Predictors of decannulation failure | 5 years
  Assessment of the presence of predictors of decannulation failure
Time of decannulation and its influence on the weaning process | 5 years
  Investigation if timing of decannulation can influence the result of the tracheostomy weaning process
Shared protocol and clinical score | 5 years
  Possible derivation of a novel clinical score and a shared protocol for decannulation

CONTACTS AND LOCATIONS:
Locations (1):
- L. Sacco Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No